CLINICAL TRIAL: NCT03803176
Title: Effect Of Periodontal Surgery On Tissue Plasminogen Activator And Plasminogen Activator Inhibitor Type-1 Gene Expression In Gingival Tissues Of Chronic Periodontitis Patients
Brief Title: Tissue Plasminogen Activator & Plasminogen Activator Inhibitor Type-1 In Gingival Tissues Of Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gihane Gharib Madkour, Associate Professor, Cairo University
Other Study IDs: 12081976
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontally healthy subjects: Healthy subjects who attended the restorative dental clinic and have clinically healthy gingiva with zero plaque index (PI), gingival index (GI), and CAL (≤3 mm PD). Oral hygeine instructions will be given to these patients.
- Chronic Periodontitis: Patients with severe Chronic Periodontitis having a pocket depth (PD) of ≥5 mm and a clinical attachment level (CAL) ≥5 mm. Open flap debridement (surgical periodontal therapy) will be carried out for these patients after scaling & root planing.
  Interventions: Procedure: Open Flap Debridement

INTERVENTIONS:
Procedure: Open Flap Debridement — Full thickness flaps are elevated to fully expose the periodontaldefects. Defects are then fully debrided and the roots are carefully planned. Flaps are repositioned and sutured to obtain primary closure of the interdental space. This will be done for chronic periodontitis patients
  Groups: Chronic Periodontitis

SUMMARY:
Tissue Plasminogen Activator and Plasminogen Activator Inhibitor Type-1 Gene Expression will be evaluated clinically and histopathologically through Hematoxylin and eosin as well as by quantitative reverse transcription polymerase chain reaction in the gingival tissues of chronic periodontitis in an attempt to investigate whether the expression of these proteins could be involved in the disease pathogenesis or not, and to assess as well if their expression will be affected by the applied surgical periodontal treatment.

DETAILED DESCRIPTION:
30 subjects were enrolled in this study and divided into: Group I (Control Group): 10 periodontally healthy volunteers, Group II (Chronic Periodontitis Group): 20 patients suffering severe CP and Group III (Treated Group): 20 patients who were scheduled for OFD. Gingival samples were collected from all subjects at baseline and at 3 months after OFD from the CP patients. Then, Hematoxylin and eosin (H&E) stained slides were examined and gene expression levels of t-PA and PAI-1 were measured in the gingiva through quantitative reverse transcription polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe chronic periodontitis
* Pocket depth (PD) of ≥5 mm
* Clinical attachment level (CAL) ≥5 mm

Exclusion Criteria:

* Pregnant women
* Subjects taking any type of medication and/or antibiotic therapy during the 3 months before the study
* Subjects who received periodontal treatment within the past 6 months
* Smokers

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population includes 30 subjects recruited from the outpatient clinic of Oral Medicine & Periodontology department, Faculty of Dentistry, Cairo University. Ages range from 30-50 years old.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 4 weeks
  CAL

CONTACTS AND LOCATIONS:
Overall Officials: Gihane G Madkour, Ass Prof, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt